CLINICAL TRIAL: NCT05791045
Title: Single Lumen Intubation and Heart-Lung Machine (HLM) Mode Ventilation Study in Endoscopic Thoracic Sympathetic Blockade
Brief Title: Single Lumen Intubation and Heart-Lung Machine (HLM) Mode Ventilation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biruni University (Other)
Responsible Party: Principal Investigator, ILKE KUPELI, Assoc. prof, Biruni University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: Biruni HLM
Record Dates: First submitted 2023-03-17; First posted 2023-03-30 (Actual); Last update posted 2023-03-30 (Actual); Status verified 2023-03

CONDITIONS: Anesthesia Time

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- double lumen tube (Active Comparator): In the DLT group, the lung on the side to be treated was distinguished from the ventilator and extinguished and single lung ventilation was performed with the other lung.
  Interventions: Procedure: single vs double
- single lumen tube (Active Comparator): In the SLT group, after thoracoscopic input, the anesthetist was in contact with the surgeon and his lung pressures were reduced manually until the lowest pressure, where the surgeon's vision was optimal.
  Interventions: Procedure: single vs double

INTERVENTIONS:
Procedure: single vs double — we aimed to compare anesthetic outcomes of single lumen intubation with Heart-Lung Machine mode ventilation versus double lumen intubation study in endoscopic thoracic sympathetic blockade

SUMMARY:
In this trial, we aimed to compare anesthetic outcomes of single lumen intubation with Heart-Lung Machine mode ventilation versus double lumen intubation study in endoscopic thoracic sympathetic blockade.

ELIGIBILITY:
Inclusion Criteria:

* 135 patients underwent bilateral ETSB procedure under general anesthesia

Exclusion Criteria:

* patients who underwent one sided ETSB
* patients under the age of 18
* Patients over 65 years of age

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-05-01 (Actual)

PRIMARY OUTCOMES:
anesthesia time | 1 year
  anesthesia time during intubation

CONTACTS AND LOCATIONS:
Locations (1):
- Ilke Kupeli, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hashmonai M, Kopelman D. History of sympathetic surgery. Clin Auton Res. 2003 Dec;13 Suppl 1:I6-9. doi: 10.1007/s10286-003-1103-5. PMID 14673664
- [Result] Caso R, Kelly CH, Marshall MB. Single lumen endotracheal intubation with carbon dioxide insufflation for lung isolation in thoracic surgery. Surg Endosc. 2019 Oct;33(10):3287-3290. doi: 10.1007/s00464-018-06614-9. Epub 2018 Dec 3. PMID 30511311